CLINICAL TRIAL: NCT05059873
Title: A Multicenter Double-blind Randomized Controlled Trial of Systemic Corticosteroid Therapy in AECOPD Patients Admitted to Hospital With Higher Blood Eosinophil Levels
Brief Title: Treatment Efficacy of Systemic Corticosteroids in AECOPD Patients With Higher Blood Eosinophil Levels
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruiting subjects
Sponsor: Capital Medical University (Other)
Collaborators: Peking University (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Xuanwu Hospital, Beijing (Other); Beijing Anzhen Hospital (Other); Beijing Tongren Hospital (Other); Beijing Luhe Hospital (Other); Emergency General Hospital (Other); Beijing Jishuitan Hospital (Other); Beijing Jingmei Group Hospital (Unknown); Bejing INFI-SAGACITY TECHNOLOGY CO., LTD (Unknown); Chinese People's Liberation Army of China General Hospital (Unknown); Beijing Yanhua Hospital (Unknown); Peking University Shougang Hospital (Other); The First Hospital of Fangshan District (Unknown); Liangxiang Hospital (Unknown); Beijing Huairou Hospital (Other)
Responsible Party: Principal Investigator, Zhaohui Tong, Derictor of Beijing Institute of Respiratory Medicine and Vice president of Beijing Chao-Yang Hospital, Capital Medical University, Beijing, China, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z201100005520029
Record Dates: First submitted 2021-09-18; First posted 2021-09-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Acute Exacerbation of COPD; Corticosteroid; Morality; Lung Diseases, Obstructive; Blood Eosinophil Count; COPD; Pulmonary Disease, Chronic Obstructive
Keywords: Treatment failure rates; Chronic Obstructive Pulmonary Disease; Randomized Controlled Trial; Mortality; Corticosteroid; Acute Exacerbation of Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic corticosteroid group (Experimental): Patients will receive Oral prednisone 40mg/day for five consecutive days in addition to standard treatment during emergency admission or hospitalization.
  Interventions: Drug: Prednisone
- Control group (Placebo Comparator): Participating patients will receive an oral placebo of 40mg/day for five consecutive days in addition to standard treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Oral prednisone 40mg/day for five consecutive days
  Arms: Systemic corticosteroid group
Drug: Placebo — Oral placebo of 40mg/day for five consecutive days
  Arms: Control group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is one of the top three causes of death worldwide now. Acute exacerbations (AEs) of COPD are a risk factor for lung function deterioration, poor quality of life, longer hospitalization, and increased mortality. To date, COPD is associated with a heavy clinical and socioeconomic burden, of which AEs of COPD account for a significant part of the cost of patients with COPD. Although several retrospective cohort studies and post-hoc analyses from randomized controlled trials (RCTs) showed that AECOPD patients with higher blood eosinophils had a shorter length of hospital stay (LOS), lower doses of corticosteroid use, and better response to systematic corticosteroid treatment than those with lower blood eosinophils, the efficacy of systematic corticosteroids in AECOPD patients with higher blood eosinophils has not been confirmed by RCTs. Therefore, this study aims to evaluate if AECOPD patients admitted to hospitals with higher blood eosinophil levels could benefit from systemic corticosteroid therapy. In this study, all eligible AECOPD participants with peripheral blood eosinophil blood count >2% or > 300 cells/μL will be randomly assigned (1:1) to either a control group or a systemic corticosteroid group. The control group will receive an oral placebo of 40mg/day for five consecutive days in addition to standard treatment during emergency admission or hospitalization. And systemic corticosteroid group will receive oral prednisone 40mg/day for five consecutive days and standard treatment. This study will provide evidence on using peripheral blood eosinophil blood count to guide corticosteroid therapy in AECOPD patients and help the clinician make an individual decision for each patient.

DETAILED DESCRIPTION:
Data about individual deidentified participants of this trial will be available from the corresponding author Zhaohui Tong (Email: tongzhaohuicy@sina.com) on reasonable request after the main results of the ECHO study have been published.

ELIGIBILITY:
Inclusion Criteria:

1. Within 24 hours of admission;
2. Aged between of 40 and 80 years old;
3. Established clinical history of COPD with spirometry-verified COPD (defined as post-bronchodilator forced expiratory volume in one second (FEV1)/ forced vital capacity (FVC) ≤ 0.70);
4. AECOPD diagnosis in accordance with the GOLD guideline (An acute worsening of respiratory symptoms that result in additional therapy)12;
5. Current or former cigarette smokers (≥10 packs per year);
6. Blood eosinophil count > 2% or >300 cells/μL tested within 24 hours of admission;
7. Signed informed consent.

Exclusion Criteria:

1. Admission due to other diseases (pneumonia, pneumothorax, pulmonary interstitial disease, active tuberculosis or bronchiectasis, ect);
2. Regular use of glucocorticoid ≥3 months;
3. Received prednisone ≥ 60 mg in the past three days (or equivalent doses of other corticosteroid);
4. Allergic or intolerant to corticosteroid;
5. Participating in or completed another drug trial within 90 days;
6. Pregnancy or lactation;
7. Severe COPD exacerbation requiring invasive mechanical ventilation (IMV) or transfer to ICU within 24 hours after emergency admission or hospitalization;
8. With complications that may cause eosinophilia;
9. Pulmonary embolism within the past two years;
10. Myocardial infarction, uncontrollable congestive heart failure or arrhythmia within the past four weeks;
11. Comorbidity that may influence the immune system;
12. Malignant tumor;
13. Neuromuscular disease affecting the respiratory system;
14. Systemic fungal infection;
15. Thoracotomy or bronchoscopic lung volume reduction surgery history;
16. Adrenocortical insufficiency history;
17. Diabetes mellitus with poor glycemic control;
18. Uncontrollable severe psychiatric illnesses even with medication, cognitive impairment, and severe language difficulties;
19. ALT ≥ 100U/L or AST ≥ 80U/L;
20. Serum creatinine ≥ 162umol/L;
21. Life expectancy of less than 30 days.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Treatment failure rates | 30 days
  Collect during index hospitalization and within 30 days after discharge. Treatment failure is defined as either one of events: a) requiring or receiving invasive or non-invasive MV during the index hospitalization; b) requiring or transferring to ICU during the index hospitalization; c) length of index hospitalization longer than 14 days; d) death during the index hospitalization or within 30 days after discharge; e) readmission with acute exacerbations of COPD within 30 days after discharge.

SECONDARY OUTCOMES:
Requiring or receiving invasive or non-invasive MV during the index hospitalization | 14 days
  Collect during index hospitalization.
Requiring or transferring to ICU during the index hospitalization | 14 days
  Collect during index hospitalization.
Length of index hospitalization longer than 14 days | 14 days
  Collect during index hospitalization.
Death during the index hospitalization or within 30 days after discharge | 30 days after discahrge
  Collect during index hospitalization and 30-day follow-up.
Readmission with acute exacerbations of COPD within 30 days after discharge | 30 days after discahrge
  Collect during index hospitalization and 30-day follow-up.
All-cause mortality within 90 days after discharge | 90 days after discahrge
  Collect during 90-day follow-up.
Readmission rates of AECOPD at 60-day and 90-day follow-ups | 90 days after discahrge
  Collect during 90-day follow-up.
Time to readmission of AECOPD within 90 days after discharge | 90 days after discharge
  Collect during 90-day follow-up.
Severer infection or development of pneumonia during hospitalization | 14 days
  Collect during index hospitalization.
Changes in the scores of Hospital Anxiety and Depression Scale between index hospitalization and 90-day follow-up | 90 days
  Collect during 90-day follow-up. The minimum and maximum values are 14 and 70, respectively. Higher scores mean a worse outcome.
Changes in the scores of St. George's Respiratory Questionnaire between index hospitalization and 90-day follow-up | 90 days
  Collect during 90-day follow-up. The minimum and maximum values are 1 and 80, respectively. Higher scores mean a worse outcome.
Changes in the scores of exacerbations of chronic pulmonary disease tool between index hospitalization and 90-day follow-up | 90 days
  Collect during huopitalization and 90-day follow-up. The minimum and maximum values are 14 and 73, respectively. Higher scores mean a worse outcome.
Changes in the scores of modified Medical Research Council Dyspnoea Scale between index hospitalization and 90-day follow-up | 90 days
  Collect during huopitalization and 90-day follow-up. The minimum and maximum values are 1 and 5, respectively. Higher scores mean a worse outcome.
Changes in the scores of COPD Assessment Test between index hospitalization and 90-day follow-up | 90 days
  Collect during huopitalization and 90-day follow-up. The minimum and maximum values are 0 and 40, respectively. Higher scores mean a worse outcome.
Changes in the scores of Transition Dyspnea Index between index hospitalization and 90-day follow-up | 90 days
  Collect during huopitalization and 90-day follow-up.
Changes in the scores of COPD Exacerbation Recognition Tool during 90-day follow-up | 90 days after discharge
  Collect during 90-day follow-up by patients.
Length of hospital stay during hospitalization | 14 days
  Collect during huopitalization

CONTACTS AND LOCATIONS:
Overall Officials: Tong Zhaohui, PhD, Study Chair — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data about individual deidentified participants of this trial will be available from the corresponding author Zhaohui Tong (Email: tongzhaohuicy@sina.com) on reasonable request after the main results of the ECHO study have been published
Supporting Information: Study Protocol, ICF
Time Frame: After the main results of the ECHO study have been published
Access Criteria: Supporting information will be available from the corresponding author Zhaohui Tong (Email: tongzhaohuicy@sina.com)

REFERENCES:
- [Background] Labaki WW, Rosenberg SR. Chronic Obstructive Pulmonary Disease. Ann Intern Med. 2020 Aug 4;173(3):ITC17-ITC32. doi: 10.7326/AITC202008040. PMID 32745458
- [Background] Duffy SP, Criner GJ. Chronic Obstructive Pulmonary Disease: Evaluation and Management. Med Clin North Am. 2019 May;103(3):453-461. doi: 10.1016/j.mcna.2018.12.005. Epub 2019 Mar 14. PMID 30955513
- [Background] Sivapalan P, Lapperre TS, Janner J, Laub RR, Moberg M, Bech CS, Eklof J, Holm FS, Armbruster K, Sivapalan P, Mosbech C, Ali AKM, Seersholm N, Wilcke JT, Brondum E, Sonne TP, Ronholt F, Andreassen HF, Ulrik CS, Vestbo J, Jensen JS. Eosinophil-guided corticosteroid therapy in patients admitted to hospital with COPD exacerbation (CORTICO-COP): a multicentre, randomised, controlled, open-label, non-inferiority trial. Lancet Respir Med. 2019 Aug;7(8):699-709. doi: 10.1016/S2213-2600(19)30176-6. Epub 2019 May 20. PMID 31122894
- [Background] Seemungal TA, Donaldson GC, Paul EA, Bestall JC, Jeffries DJ, Wedzicha JA. Effect of exacerbation on quality of life in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 May;157(5 Pt 1):1418-22. doi: 10.1164/ajrccm.157.5.9709032. PMID 9603117
- [Background] Wedzicha JA, Singh R, Mackay AJ. Acute COPD exacerbations. Clin Chest Med. 2014 Mar;35(1):157-63. doi: 10.1016/j.ccm.2013.11.001. PMID 24507843
- [Background] Bafadhel M, Greening NJ, Harvey-Dunstan TC, Williams JE, Morgan MD, Brightling CE, Hussain SF, Pavord ID, Singh SJ, Steiner MC. Blood Eosinophils and Outcomes in Severe Hospitalized Exacerbations of COPD. Chest. 2016 Aug;150(2):320-8. doi: 10.1016/j.chest.2016.01.026. Epub 2016 Feb 3. PMID 26851799
- [Background] Cui Y, Zhan Z, Zeng Z, Huang K, Liang C, Mao X, Zhang Y, Ren X, Yang T, Chen Y. Blood Eosinophils and Clinical Outcomes in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease: A Propensity Score Matching Analysis of Real-World Data in China. Front Med (Lausanne). 2021 Jun 9;8:653777. doi: 10.3389/fmed.2021.653777. eCollection 2021. PMID 34179040
- [Background] Ko FWS, Chan KP, Ngai J, Ng SS, Yip WH, Ip A, Chan TO, Hui DSC. Blood eosinophil count as a predictor of hospital length of stay in COPD exacerbations. Respirology. 2020 Mar;25(3):259-266. doi: 10.1111/resp.13660. Epub 2019 Aug 6. PMID 31385389
- [Derived] Liang L, Lin Y, Feng L, Shao S, Cao S, Rong H, Chu S, Xie W, Cai S, Wang J, Tong Z. Multicentre double-blind randomised controlled trial of systematic corticosteroid therapy in patients with acute exacerbations of chronic obstructive pulmonary disease admitted to hospital with higher eosinophil levels: the ECHO protocol. BMJ Open. 2023 May 29;13(5):e066354. doi: 10.1136/bmjopen-2022-066354. PMID 37247957
- See also: Chinese expert consensus on the diagnosis and treatment of acute exacerbation of chronic obstructive pulmonary disease (AECOPD) (updated version in 2017) — http://rs.yiigle.com/CN131368201714/1000344.htm